CLINICAL TRIAL: NCT05520294
Title: Evaluating the Effects of Cannabis Use and Circulating Cannabinoids on Tumor Infiltrating Lymphocytes in Malignant Melanoma
Status: Active, not recruiting | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Collaborators: Cancer League of Colorado (Other)
Responsible Party: Sponsor
Other Study IDs: 22-1132
Record Dates: First submitted 2022-08-25; First posted 2022-08-29 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Paraffin Tissue Blocks Whole Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Chronic Cannabinoid Users: Ib or II Melanoma patients who are chronic cannabinoid users
  Interventions: Other: High-performance liquid chromatography-tandem mass spectrometry assays
- Non-users: Ib or II Melanoma patients non cannabinoid users
  Interventions: Other: High-performance liquid chromatography-tandem mass spectrometry assays

INTERVENTIONS:
Other: High-performance liquid chromatography-tandem mass spectrometry assays — Paraffin blocks will be requested for slide creation, and at least 12 mL of whole blood will be collected in 2 green top tubes, centrifuged, and plasma transferred for storage at -80 C until further processing

SUMMARY:
The goal of this proposal is to determine how cannabinoid use affects the tumor immune microenvironment (TME) of melanoma by correlating TILs with reported cannabinoid use and circulating plasma cannabinoids. The central hypothesis is that cannabinoid use decreases TILs in melanoma in a dose-dependent fashion. This is important because cannabinoid-driven TME changes in melanoma may alter patient outcomes mediated by TILs and response to standard of care ICI treatments.

DETAILED DESCRIPTION:
Specific Aim 1.Assess how systemic cannabinoids remodel tumor infiltrating lymphocytes (TILs) within the melanoma tumor microenvironment. We hypothesize that decreased grade of TILs and exhaustive differentiation of T cells in melanoma are associated with lower cannabinoid receptor (CB1/CB2) expression and higher levels of systemic exogenous cannabinoids. Aim 1a.) Correlate plasma levels of cannabinoids with TIL grade. Aim 1b.) Correlate plasma levels of cannabinoids with TIL T cell immunohistochemical markers of exhaustion. Aim 1c.) Correlate plasma levels of cannabinoids to TIL CB1/CB2 expression.

Specific Aim 2. Determine the relationship between peripheral T cell activation and circulating cannabinoid levels in patients with melanoma. We hypothesize that the phenotypic activation of peripheral T cells is inversely associated with increased plasma levels of systemic exogenous cannabinoids. Aim 2a.) Immunophenotype peripheral T cells from patients with melanoma. Aim 2b.) Correlate plasma levels of cannabinoids with peripheral T cell phenotypic activation.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy proven melanoma, any stage

  * Biopsy obtained within 4 weeks of anticipated enrollment
  * Patients >21 years old
  * Report no cannabis use in the last year or chronic cannabis use (at least weekly use for 3 months or more)

Exclusion Criteria:

* Patients unwilling or unable to provide informed consent

Ages: 21 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Description of Population to be Enrolled:
  Patients who are either chronic cannabis/cannabinoid users (use >1 time/week for >3 months of any cannabinoid product, with ingestion via edibles, smoking, or vaping) and non-users for the last year who are scheduled to be seen in a clinic at the University of Colorado Cancer Center will be approached for enrollment and informed consent. Enrollment will be limited to stage Ib and II to decrease patient heterogeneity and since higher TIL grade has been associated with earlier stage melanomas13, thus maximizing the potential to observe an effect. Biopsy specimens must be obtained within 4 weeks of study enrollment to ensure blood specimens are reflective of when biopsy specimens were obtained.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2024-08-31 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Grade of TIL in melanoma biopsy | 24 Months
  Hematoxylin and eosin slide assessment
Composition of TILs within melanoma biopsy specimens | 24 Months
  Stains for TIL markers such as CD3, CD4, CD8, CD20, CD45RO, and FoxP3; T cell function IHC stains include: TOX, PD1, TIGIT, LAG3; melanoma specific marker SOX10

CONTACTS AND LOCATIONS:
Overall Officials: Camille Stewart, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Denver, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: Undecided